CLINICAL TRIAL: NCT06020196
Title: The Safety and Efficacy of Surgical Rectus Sheath Block Compared to Subdermal Infiltration of Local Anaesthetic for Postoperative Analgesia After Elective Cesarean Section: a Randomized Control Trial
Brief Title: The Safety and Efficacy of Surgical Rectus Sheath Block for Postoperative Analgesia After Elective Cesarean Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ahmed M Maged, MD (Other)
Responsible Party: Sponsor-Investigator, Ahmed M Maged, MD, Professor of Obstetrics and Gynecology at Cairo University, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 71
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Post Operative Pain
Keywords: surgical rectus sheath block; sudermal infiltration of local anaesthesia; cesarean section
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This study will be a prospective, single-blinded, randomized controlled trial (RCT) that include 182 patients scheduled for an elective lower segment Cesarean section at the Obstetrics and Gynecology department of Kasr Alainy University Hospital from April 2023 to August 2023.
  After obtaining approval from the hospital's institutional review board, we assessed 182 young women scheduled for an elective lower segment Cesarean section to determine their eligibility for the study.
  The182 patients admitted to be enrolled in our study, in which they're randomized into 2 groups, Group 1(n= 91) received bilateral surgical rectus sheath block and Group 2 (n =91) received subdermal infiltration of local anaesthetics.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rectus sheath block group (Active Comparator): The participants will receive bilateral surgical rectus sheath block
  Interventions: Procedure: surgical rectus sheath block
- Subdermal group (Active Comparator): The participants will receive subdermal infiltration of local anaesthetics.
  Interventions: Procedure: subdermal local anaesthetic infiltration

INTERVENTIONS:
Procedure: surgical rectus sheath block — Local anaesthetic will be administered into the rectus sheath space by the surgeon, towards the end of the operation, at the time of closure of the anterior abdominal wall (before the closure of peritoneum)
  Arms: Rectus sheath block group
Procedure: subdermal local anaesthetic infiltration — After closure of the subcutaneous fat, the edges of the skin become more stable; subdermal Infiltration with moving needle technique was done to optimize distribution of the local anesthetic solution
  Arms: Subdermal group

SUMMARY:
All participants will receive spinal anaesthesia and will be randomly divided into 2 equal groups. In Group 1, 20 ml of local anesthetic solution will be administered bilaterally to the rectus sheath space under direct vision before closure of the anterior abdominal wall. Meanwhile, Group II will receive subdermal injections of 20 ml of local anesthetic solution before closure of the skin. Each 20 ml of local anaesthetic solution contained 0.25% Bupivacaine (50 mg/ 20 ml), 4mg dexamethazone and 1:200,000 epinephrine.

DETAILED DESCRIPTION:
All participants will receive spinal anaesthesia and will be randomly divided into 2 equal groups. In Group 1, 20 ml of local anesthetic solution will be administered bilaterally to the rectus sheath space under direct vision before closure of the anterior abdominal wall. Meanwhile, Group II will receive subdermal injections of 20 ml of local anesthetic solution before closure of the skin. Each 20 ml of local anaesthetic solution contained 0.25% Bupivacaine (50 mg/ 20 ml), 4mg dexamethazone and 1:200,000 epinephrine.

All cases will be followed up hourly for 6 hours postoperative for assessment of level of pain by using visual analog scale (VAS). Primary outcome parameters were VAS score during rest and the need for additional analgesics during the first 48 post-operative hours. Other parameters will be time of start of lactation and ambulation, length of post-operative hospital stay, and occurrence of side effects or complications.

ELIGIBILITY:
Inclusion Criteria:

* Women with singleton pregnancies.
* Gestational age 37 to 41 weeks.
* Surgical history: no history of previous surgeries or history of previous 1 cesarean section,
* Age: 20 -35 years old,
* American Society of Anesthesiologists physical status classifications II (healthy pregnancy or with mild systemic disease) [Amr E. Abouleish et. al. 2015],
* Scheduled for elective cesarean section
* BMI: 18.5 - 35 kg/m2.

Exclusion Criteria:

* if they had American Society of Anaesthesiologists (ASA) status III and above (with severe systemic disease),
* Patients with BMI < 18.5 or > 35 kg/m2 were excluded as they require a different dosage of drug for spinal anesthesia,
* History of previous 2 Caesarian or more,
* Known allergy to the drug used (bupivacaine),
* Contraindication to NSAID: patients with suspected or manifest bleeding disturbances, allergy to NSAID, atopia, bronchial asthma, diabetes mellitus, those who previously had shown marked side effects after NSAID, the presence of liver or kidney disease, abuse of drugs or alcohol, excessive smokers and patients with pregnancy induced hypertension or pre-eclampsia
* Bleeding disorders, e.g.: thrombocytopenia,
* Neurological disorders associated with sensory alterations, e.g., Transverse myelitis can cause back pain, abnormal sensations in the trunk and genital region and legs such as sensory loss or paresthesias (abnormal sensations such as burning, tickling, pricking, numbness, coldness, or tingling).
* Rheumatological diseases e.g., primary Sjögren's syndrome (pSS), systemic lupus erythematosus (SLE) and rheumatoid arthritis (RA), accompanied by chronic widespread pain due to arthralgia, myalgia or serositis.
* Requiring general anesthesia,
* if vertical abdominal incision was required,
* Local infection at the site of injection or
* The inability to provide a pain score, e.g., visual impairement.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 182 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
postoperative pain during rest | 6 hours
  All cases will be followed up hourly for 6 hours postoperative for assessment of level of pain by using visual analog scale (VAS)
the amount of additional analgesics consumption post-operatively for pain relief. | 48 hours
  assessment amount of intravenous analgesic consumption during hospital stay. Also, an investigator contacted them 24 hours after discharge to monitor oral analgesic analgesic

SECONDARY OUTCOMES:
time of start of lactation | 24 hours
  the interval between skin closure and the time the patient first breastfeeds her newborn.
time of start of ambulation | 24 hours
  the interval between skin closure and the time patient first ambulated.
length of post-operative hospital stay | 24 hours
  the interval between skin closure and the time patient discharged from hospital.
development of of side effects or complications. | 24 hours
  The patient was observed for potential complications of RSB:
  The superior and inferior epigastric arteries are at risk of injury Visceral damage, Local anesthetic systemic toxicity, leading to seizures or ventricular arrhythmias (rare) Incomplete block may result from anatomical variance, as in up to 30% of the population.
  Failure of the block as the posterior wall of the rectus sheath lying superficial to the peritoneal cavity, needle misplacement may lead to injection into the peritoneal cavity.
  Infection.
  The patient was observed for potential complications of subdermal local anesthetic infilteration, including wound infection
  also the paients were observed for developemt of NSAID side effec

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M. Maged, Professor, Study Chair — Professor of Obstetrics and Gynecology at Cairo University
Locations (1):
- The Obstetrics and Gynecology department of Kasr Alainy University Hospital, Cairo, El Manial, Egypt

IPD SHARING:
Plan to Share IPD: No